CLINICAL TRIAL: NCT02972593
Title: ORthopaedic Trauma Anemia With Conservative Versus Liberal Transfusion
Acronym: ORACL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Atlanta Medical Center (Other)
Responsible Party: Principal Investigator, Brian Mullis, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1402557771
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Blood Specimen Collection; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal (Other): Blood and blood products for transfusion. Transfusion will be done to keep Hgb >7 g/dL.
  Interventions: Biological: Blood and blood products for transfusion
- Conservative (Other): Blood and blood products for transfusion. Transfusion will be done to keep Hgb > 5.5 g/dL.
  Interventions: Biological: Blood and blood products for transfusion

INTERVENTIONS:
Biological: Blood and blood products for transfusion — Randomization would not occur until the patient's Hgb dropped below 7 g/dL. If the patient is randomized to the liberal arm, they would be transfused to keep their Hgb >7 g/dL. If the patient is randomized to the conservative arm, they would not be transfused until their Hgb drops below 5.5 g/dL. If the patient's Hgb does not drop below 7.0 g/dL, randomization will not be done.

SUMMARY:
The purpose of this study is to determine if there is a difference in outcomes between liberal transfusion (transfusing when hemoglobin drops below a set higher value number) and conservative transfusion (transfusing when hemoglobin drops below a set lower value number).

DETAILED DESCRIPTION:
Transfusion of Orthopaedic trauma patients is routinely done in asymptomatic individuals as there is no accepted national standard or recommendations from the American Academy of Orthopaedic Surgeons or the Orthopaedic Trauma Association for what level of anemia is appropriate in an asymptomatic patient. Individual practitioners typically make this decision based on anecdotal experiences and expert opinion. No prospective study has been performed to date to answer this question in this patient population.

The null hypothesis of this proposed pilot study is that no difference will be seen with a liberal transfusion strategy to keep a patient's hemoglobin above 7 g/dL versus a conservative strategy to keep the patient's hemoglobin above 5.5 g/dL in patients asymptomatic at rest. The primary outcome of this pilot study will be infection; defined as postoperative wound infection (superficial or deep) or other perioperative infection but not surgical site (urinary tract infection or pneumonia). Deep infection is defined as the need for intravenous antibiotics or a return to surgery for debridement. Superficial infection is defined as the use of oral antibiotics only successfully treat a surgical site infection. Secondary outcomes will include pulmonary embolism, deep venous thrombosis, acute renal failure or insufficiency, nonunion, delayed union, compartment syndrome, osteomyelitis, nerve palsy, anoxic brain injury, cardiac ischemia or infarct, pancreatitis, or death, and the musculoskeletal functional assessment.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients admitted to participating hospital with any Orthopaedic injury who have been determined to be stable by the Trauma Service (General Surgery) and are no longer within the resuscitation phase of initial treatment. This is defined as a normal urine output (greater than 0.5 ml/kg/hr) and a systolic blood pressure greater than 90 mmHg for greater than 6 hours without fluid bolus or transfusion during that time
* Age 18-50
* Hemoglobin less than 9 g/dL or expected drop below 9 g/dL with planned surgery

Exclusion Criteria:

* Pregnant ( urine pregnancy test will be done as standard of care)
* Prisoner
* Head injury (Glasgow Coma Scale less than 8 over 48 hours from presentation)
* Known cardiac (coronary artery disease, atrial fibrillation, stent placement, congestive heart failure), renal (acute or chronic renal insufficiency or failure, defined as having Serum Creatinine >1.2 at time of enrollment), liver (Childs C cirrhosis) or pulmonary disease (chronic obstructive pulmonary disease, abnormal pulmonary function tests or history of poor pulmonary function from any cause including acute traumatic conditions such as ARDS)
* Unlikely to follow up in the surgeon's estimation
* Sickle Cell Anemia
* History of cancer
* Preexisting weakness, paresthesias, deformities, or other conditions which might affect functional outcome in the surgeon's opinion
* Spinal cord injury
* Patients with burns expected to require operative treatment
* COVID positive

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian H Mullis, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mullis BH, Mullis LS, Kempton LB, Virkus W, Slaven JE, Bruggers J. Early Results of Orthopaedic Trauma and Anemia: Conservative Versus Liberal Transfusion Strategy. J Am Acad Orthop Surg. 2024 Mar 1;32(5):228-235. doi: 10.5435/JAAOS-D-23-00235. Epub 2023 Dec 27. PMID 38154083
- [Derived] Mullis BH, Mullis LS, Kempton LB, Virkus W, Slaven JE, Bruggers J. Orthopaedic Trauma and Anemia: Conservative versus Liberal Transfusion Strategy: A Prospective Randomized Study. J Orthop Trauma. 2024 Jan 1;38(1):18-24. doi: 10.1097/BOT.0000000000002696. PMID 38093439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 3 level 1 trauma centers between March 2014 and May 2021. The first patient was enrolled on March 11, 2014 and the last participant was enrolled on May 7, 2021.
Pre-assignment Details: Screening/IC done on 161 patients with a Hgb of ≤9g/dL or whose Hgb was expected to drop below 9g/dL with planned procedures/continued (controlled) bleeding. Randomization assignment occurred once patient's Hgb dropped below 7g/dL. Out of the 161 patient that consented, there were 61 whose Hgb did not drop below 7g/dL and randomization was not performed on. Those 61 patients were considered screen failures, leaving 100 patients who were randomized to either liberal or conservative transfusion.
Groups:
- Liberal: Blood and blood products for transfusion. Transfusion will be done to keep Hgb >7 g/dL.
  Blood and blood products for transfusion: Randomization would not occur until the patient's Hgb dropped below 7 g/dL. If the patient is randomized to the liberal arm, they would be transfused to keep their Hgb >7 g/dL.
- Conservative: Blood and blood products for transfusion. Transfusion will be done to keep Hgb > 5.5 g/dL.
  If the patient is randomized to the conservative arm, they would not be transfused until their Hgb drops below 5.5 g/dL.
Period: Overall Study
Arm/Group | Liberal | Conservative
Started | 50 | 50
Completed | 30 | 35
Not Completed | 20 | 15
Not completed — Lost to Follow-up | 19 | 15
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: One hundred patients were enrolled and randomized; however, it was noted the day after enrollment for a patient in the liberal group that the patient should not have been enrolled due to a creatinine higher than allowed by the exclusion criteria. The patient was immediately removed from the study and not included in the statistical analysis.
Groups:
- Liberal Transfusion: Transfusion will be done to keep Hgb >7 g/dL.
- Conservative Transfusion: Transfusion will be done to keep Hgb > 5.5 g/dL.
- Total: Total of all reporting groups
Arm/Group | Liberal Transfusion | Conservative Transfusion | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 50 | 99
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 45 | 4 | 49
  Unknown or Not Reported | 2 | 41 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 18 | 38
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Wound Infection (Superficial or Deep) or Other Perioperative Infection
Description: Deep infection is defined as the need for intravenous antibiotics and/or a return to surgery for debridement. Superficial infection is defined as clinical diagnosis of cellulitis or other superficial infection treated with oral antibiotics only.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Groups:
- Liberal: Transfusion will be done to keep Hgb >7 g/dL.
- Conservative: Transfusion will be done to keep Hgb > 5.5 g/dL.
Arm/Group | Liberal | Conservative
Number analyzed (Participants) | 49 | 50
Participants | 12 | 3
Statistical Analysis 1: Comparison: Liberal vs Conservative; Test type: Other — Data collapsed to participant level, creating an ever/never response for each participant for each infection outcome type. Analyses performed at the participant level to determine if proportion of outcome types were similar between transfusion groups using Fisher's Exact tests, due to small expected cell counts, using SAS v9.4 (SAS Institute, Cary, NC). Power analyses performed based on these proportions using bootstrapping methods in SAS and confirmed with nQuery v8.7.1.0; p = .0122, Fisher Exact

2. Secondary Outcome: Combined Secondary Outcomes
Description: Combined (any) Secondary Outcomes: pulmonary embolism, deep venous thrombosis, acute renal failure or insufficiency, nonunion, delayed union, compartment syndrome, osteomyelitis, nerve palsy, anoxic brain injury, cardiac ischemia or infarct, pancreatitis, or death.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Groups:
- Liberal: Transfusion will be done to keep Hgb >7 g/dL.
  Blood and blood products for transfusion: Randomization would not occur until the patient's Hgb dropped below 7 g/dL. If the patient is randomized to the liberal arm, they would be transfused to keep their Hgb >7 g/dL.
- Conservative: Transfusion will be done to keep Hgb > 5.5 g/dL.
  If the patient is randomized to the conservative arm, they would not be transfused until their Hgb drops below 5.5 g/dL.
Arm/Group | Liberal | Conservative
Number analyzed (Participants) | 49 | 50
Participants | 7 | 6
Statistical Analysis 1: Comparison: Liberal vs Conservative; Test type: Other; p = .7742, Fisher Exact

3. Secondary Outcome: Musculoskeletal Function Assessment
Description: The Musculoskeletal Function Assessment (MFA) evaluates the health status of patients with musculoskeletal disorders of the extremities, including patients with fractures and soft tissue injuries, repetitive motion disorders, osteoarthritis or rheumatoid arthritis. It describes patient functioning, assesses outcomes of surgical interventions and clinical trials, and monitors patients' functional status over time. The MFA is scored from 0 to 100 with 0 representing no dysfunction. Higher MFA scores/values represent a higher levels of dysfunction or worse outcome.
Time Frame: one year
Population: Sixty five patients completed 1 year follow up but 5 declined to complete the MFA, leaving sixty patients that completed 1 year MFA.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liberal | Conservative
Number analyzed (Participants) | 29 | 31
score on a scale | 35.9 (21.1) | 28.2 (19.4)
Statistical Analysis 1: Comparison: Liberal vs Conservative; Test type: Other; p = .1443, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Liberal | Conservative
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 7/49 | 6/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal (N=49) | Conservative (N=50)
Secondary DVT (Vascular disorders) | 2 (2) | 1 (1)
Transfusion-related acute lung injury (TRALI) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)

LIMITATIONS AND CAVEATS:
Significant loss to follow up; Significant resistance by multiple providers at each site to allow conservative treatment algorithm (as most felt liberal was standard of care); Slow enrollment; No funding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT02972593/Prot_SAP_000.pdf